CLINICAL TRIAL: NCT03048253
Title: Recombinant Human GM-CSF Herpes Simplex Virus Injection (OrienX010) Standard Injection in Tumor Treatment Scheme Failed M1c Ⅳ Period Malignant Melanoma Spread to the Liver Open I-c Phase of Clinical Trial
Brief Title: A Phase I-c Study of Recombinant GM-CSF Herpes Simplex Virus to TreatⅣ M1c
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: OrienGene Biotechnology Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: OrienX010-II-10
Record Dates: First submitted 2017-02-03; First posted 2017-02-09 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: OrienX010 — Beijing biological technology co., LTD. Research and development of the source and force of recombinant human GM-CSF herpes simplex virus injection (OrienX010), is a genetically engineered type 1 herpes simplex virus (HSV - 1) as the carrier insert GM-CSF gene therapy drug.Its carrier is made of isolated from patients with oral Chinese wild single blister virus type I (CL1), after gene recombination technology successively removing ICP34.5, ICP47 and insert the deactivation ICP6 gene, and at the site of the original ICP34.5 insert guided by IE promoter of hCMV human GM-CSF gene.

SUMMARY:
Recombinant human GM-CSF herpes simplex virus injection (OrienX010) is a genetically engineered from Chinese patients oral separation of wild type 1 herpes simplex virus (HSV) as the carrier insert GM-CSF gene therapy drug.After gene recombination technology successively removing ICP34.5, ICP47 and insert the deactivation ICP6 gene, and at the site of the original ICP34.5 insert guided by IE promoter of hCMV human gm-csf gene.The drug after tumor site local injections of dosing, on the one hand, because of the soluble tumor characteristics of herpes simplex virus, reconstructing it after HSV-1 virus carrier at the injection site specific "soluble tumor" kill tumor cells;Viral vector expressed in tumor site, on the other hand, to produce high concentrations of GM-CSF enhance the antitumor immune function, play "beside the destruction effect", have inhibition effect on the distant metastases.

DETAILED DESCRIPTION:
Subjects were tested drugs within 8 x 107 pfu/ml tumor injection treatment, the injection quantity according to tumor lesion size, injection amount shall not exceed 10 ml each time, injection frequency for every 2 weeks, 4 times per cycle treatment, treatment 2 cycles. Completed at the end of the second cycle after curative effect evaluation, such as the researchers determine continue to medicine can bring benefit to the subjects, can continue to offer benefits to the subjects' potential drug until disease progression, smaller, not tolerance toxicity or participants to withdraw consent.

ELIGIBILITY:
Inclusion Criteria:

* By histological and/or cytology diagnosis Ⅳ M1c malignant melanoma patients with liver metastasis, the lack of an effective method for the conventional or the failure of conventional therapy or recurrence
* General physical status score (ECOG) 0-2 points
* Lifetime is expected to more than 4 months
* Always anti-tumor treatment (including/radiation therapy, immune therapy, targeted therapy, endocrine therapy, etc.) to end more than 4 weeks (using the nitroso urea class and mitomycin chemotherapy drug withdrawal over 6 weeks), and always treat the adverse reaction of restored or stability

Exclusion Criteria:

* In the group treated with other experimental drugs within 4 weeks before, but in the intervening clinical research (except such as epidemiological studies)
* In group of four weeks before received the treatment of herpes simplex virus, such as acyclovir, ganciclovir, respectively.there is galloway, vidarabine, etc
* In group of four weeks before too much surgery
* Screening stage HSV - 1 antibody IgG and IgM are negative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Melanoma Standard solution phase failure Ⅳ M1c malignant melanoma spread to the liver
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-03-29 (Actual); Primary Completion 2017-10-10 (Estimated); Study Completion 2019-10-28 (Estimated)

PRIMARY OUTCOMES:
change of tumor size | 16 weeks
  According to RECIST1.1 method to evaluate the change of tumor size.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing cancer hospital, Beijing, Beijing Municipality, China